CLINICAL TRIAL: NCT03768973
Title: Pulmonary Effects of Diabetes Mellitus in Anesthetized Mechanically Ventilated Patients
Brief Title: Pulmonary Effects of Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Szeged University (Other)
Collaborators: Hungarian Basic Research Council (Other); GINOP (Unknown)
Responsible Party: Principal Investigator, Barna Babik, Professor, Szeged University
Other Study IDs: WHO2788-a
Record Dates: First submitted 2018-11-29; First posted 2018-12-07 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus; Cardiac Surgical Procedures; Respiratory Mechanics; Capnography
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group T2DM: Patients with diabetes mellitus undergoing elective cardiac surgery
  Interventions: Procedure: Elective cardiac surgery
- Group Ctrl: Control patients undergoing elective cardiac surgery without T2DM
  Interventions: Procedure: Elective cardiac surgery

INTERVENTIONS:
Procedure: Elective cardiac surgery — Both groups will undergo elective cardiac surgery as an intervention.

SUMMARY:
Type 2 diabetes mellitus (T2DM) poses a significant burden on the patients and the health care system. The increasing number of surgery performed in elderly population results in an increased number of perioperative T2DM-related adverse effects. T2DM has a prevalence of 30-40% in a population undergoing cardiovascular surgery. Cardiac surgery, especially cardiopulmonary bypass (CPB) is also known to deteriorate respiratory mechanics. The vascular effects of T2DM are well characterized, however, its effects on the mechanical properties of the respiratory system or the exhaled carbon-dioxide concentration curve (capnogram) during and following CPB are yet to be fully discovered.

Therefore, the study is aimed at characterizing the respiratory consequences of T2DM, i.e.: i: deteriorations of airway function that might be a result of smooth muscle dysfunction; ii: deterioration of the viscoelastic properties of the lung as a result of lung volume loss or structural changes, iii: exploring whether the changes of respiratory mechanics caused by cardiac surgery exhibit a different time course in T2DM and control patients.

The study also aims at characterizing the effects of T2DM on capnogram parameters: i: whether it influences capnogram shape factors, ii: whether any differences can be detected in the dead-space parameters and iii: whether cardiac surgery has a different effect on capnogram parameters in T2DM patients compared to controls.

DETAILED DESCRIPTION:
One hour before the surgery, patients are premedicated with lorazepam (per os, 2.5 mg). Induction of anaesthesia is achieved by iv midazolam (30 μg/kg), sufentanyl (0.4-0.5 μg/kg), and propofol (0.3-0.5 mg/kg), and iv propofol (50 mg/kg/min) is administered to maintain anaesthesia. Intravenous boluses of rocuronium (0.6 mg/kg for induction and 0.2 mg/kg every 30 minutes for maintenance) is administered iv to ensure neuromuscular blockade. A cuffed tracheal tube (internal diameter of 7, 8, or 9 mm) is used for tracheal intubation, and patients are mechanically ventilated (Dräger Zeus, Lübeck, Germany) in volume-controlled mode with decelerating flow. A tidal volume of 7 ml/kg and a positive end-expiratory pressure of 4 cmH2O are applied, and the ventilation frequency is adjusted to 12-14 breaths/min to maintain end-tidal CO2 partial pressure of 36 38 mmHg. Mechanical ventilation is performed with a fraction of inspired oxygen of 0.5 before CPB, and it is increased to 0.8 after CPB. As a standard part of the cardiac anaesthesia procedure, oesophageal and rectal temperature probes are introduced, and a central venous line is inserted into the right jugular vein. The left radial artery is also cannulated to monitor systolic, diastolic and mean arterial (MAP) blood pressures and arterial blood gas samples.

The membrane oxygenator is primed with 1,500 ml lactated Ringer's solution prior to CPB. Intravenous heparin (300 U/kg) is injected into the patient, to achieve an activated clotting time of 400 s during CPB procedures. During CPB, mild hypothermia is allowed, the mechanical ventilation is stopped, and the ventilator is disconnected without applying positive airway pressure. Before restoring ventilation, the lungs are inflated 3-5 times to a peak airway pressure of 30 cmH2O to facilitate lung recruitment.

A flow meter and a mainstream capnometer is to be inserted into the breathing circuit between the endotracheal tube and the Y-piece of the breathing circuit to record capnogram curves. a T-piece with 2 collapsible segments is attached to the distal tracheal tube, with one end connected to the respirator and the other end to a loudspeaker-in-box system (FOT system) to measure respiratory mechanics by the use of forced oscillations. During normal ventilation the FOT system is not communicating with the patient, however, during measurements of respiratory mechanics the ventilator is to be stopped at end-expiration and the breathing circuit is blocked in a way that allows a connection between the FOT system and the patient. During a 15-s long apnoeic period respiratory mechanical parameters are to be measured with the FOT system and then normal ventilation is to be restored. Capnogram curves are going to be recorded and respiratory mechanical parameters are going to be measured a) after anaesthesia induction with the chest wall still intact, b) following chest wall opening before CPB initiation, c) following CPB with the chest wall open and d) following sternal closure before end of surgery in all groups of patients. Arterial and venous blood gas samples are also going to be collected at these time points.

Sample sizes are estimated to enable the detection of a 15% difference in the primary outcome parameter, the lung tissue elastance. Accordingly, sample-size estimation based on an ANOVA test with two groups of patients indicated that 155 patients were required in each group to detect a significant difference between the protocol groups (the assumed variability of 30%, power of 80% and the significance level of 5%).

Two-way repeated measures ANOVA with the inclusion of an interaction term is used for all measured variables with the protocol stage as within-subject factor (protocol stages) and group allocation as between-subject factor to establish the effects of T2DM and the surgical procedure on the measured respiratory mechanical and capnography indices. At half-way of the data collection, an interim analyses will be performed and the further data collection will be proceeded based on the results of this analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery with or without diabetes mellitus
* age between 18-80 years

Exclusion Criteria:

* patients older than 80 years of age or younger than 18 years
* poor ejection fraction (<40%)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients enrolled at the Second Department of Internal Medicine and Cardiology Centre Cardiac Surgical Unit, University of Szeged
Sampling Method: Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Changes in lung input impedance and mechanical parameters | Intraoperative interval during cardiac surgery starting from anaesthesia induction until end of the surgery. (approx. 180 minutes, measurements at ~10-40-140-160 minutes)
  Changes in the airway and tissue mechanical properties are assessed by measuring the input impedance of the lungs. Briefly, a T-piece with 2 collapsible segments is attached to the tracheal tube, with one end connected to the respirator and the other to a loudspeaker-in-box system. This makes it possible to switch the patient from the respirator to the forced oscillatory setup during the measurements. The measurements are performed by introducing pseudorandom pressure excitations generated by the loudspeaker into the trachea during short (15s) apnoeic pauses introduced into the mechanical ventilation. Lung input impedance is computed from the power spectra of airway opening pressure and tracheal airflow and then averaged under each condition.
  The measured lung impedance data are fitted using a 4-element model consisting of a frequency-independent airway resistance and inertance and a constant-phase tissue compartment characterized by the coefficients of damping and elastance.
Changes of exhaled CO2 partial pressure curve shape factors | Intraoperative interval during cardiac surgery starting from anaesthesia induction until end of the surgery. (approx. 180 minutes, measurements at ~10-40-140-160 minutes)
  Changes in CO2 partial pressure in the exhaled gas during mechanical ventilation are measured with a calibrated mainstream capnograph (Capnogard Model 1265, Novametrix). A 28-mm internal diameter screen pneumotachograph connected to a differential pressure transducer (ICS model 33NA002D; IC Sensors) is used to measure airflow. The measured signals are digitized and stored on a computer. A custom-made software is used to determine parameters of this curve. The exhaled CO2 partial pressure is expressed both as a function of time (time domain) and as a function of exhaled volume (volumetric domain). Shape factors and dead-space indices of the recorded CO2 partial pressure curves are to be determined both from time and volumetric domains.
Changes in intrapulmonary shunt fraction | : Intraoperative interval during cardiac surgery starting from anaesthesia induction until end of the surgery. (approx. 180 minutes, measurements at ~10-40-140-160 minutes)
  To measure intrapulmonary shunt fraction, arterial and central venous blood gas samples are going to be obtained. The partial pressure of oxygen and carbon-dioxide in these blood samples is to be determined alongside pH and ion concentrations by radiometric blood gas analysis. Intrapulmonary shunt fraction is going to be calculated from the oxygen content of these arterial and central venous blood samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology Centre Cardiac Surgical Unit and Second Department of Internal Medicine, University of Szeged, Szeged, Csongrád megye, Hungary

IPD SHARING:
Plan to Share IPD: Undecided